CLINICAL TRIAL: NCT03472638
Title: Efficacy Of Repetitive Transcranial Magnetic Stimulation In The Treatment Of Refractory Depression Among Patients With Borderline Personality Disorder
Brief Title: Dorsomedial rTMS For Depression In Borderline Personality Disorder
Acronym: rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jonathan Downar, Director, MRI-Guided rTMS Clinic, University Health Network, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-9928
Record Dates: First submitted 2018-03-07; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Borderline Personality Disorder; Major Depression
MeSH Terms: conditions — Borderline Personality Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active -> Sham (Experimental): 15 days of active, followed by 15 days of sham rTMS, targeting dorsomedial prefrontal cortex bilaterally, two sessions per day (1 hour apart), 20 Hz stimulation, at 120% resting motor threshold
  Interventions: Device: Dorsomedial prefrontal rTMS
- Sham -> Active (Experimental): 15 days of sham, followed by 15 days of active rTMS, targeting dorsomedial prefrontal cortex bilaterally, two sessions per day (1 hour apart), 20 Hz stimulation, at 120% resting motor threshold
  Interventions: Device: Dorsomedial prefrontal rTMS

INTERVENTIONS:
Device: Dorsomedial prefrontal rTMS — Active or sham rTMS targeting the dorsomedial prefrontal cortex, 20 Hz stimulation, 120% resting motor threshold, 1500 pulses per hemisphere, using a MagVenture R30 stimulator and Cool-DB80 coil.
  Other Names: DMPFC-rTMS

SUMMARY:
This randomized trial with a crossover design will examine the efficacy of rTMS targeting the dorsomedial prefrontal cortex as a treatment for medication-resistant major depression in patients meeting diagnostic criteria for borderline personality disorder.

DETAILED DESCRIPTION:
Patients meeting standard DSM-5 diagnostic criteria for borderline personality disorder, who also meet diagnostic criteria for a major depressive episode that has not responded to medication, will be eligible for inclusion. In a study with a randomized crossover design, they will undergo a course of either either active followed by sham or sham followed by active treatment. Each phase (active or sham) will involve 15 days of rTMS targeting the bilateral dorsomedial prefrontal cortex, 5x weekly, twice-daily with sessions 1 hour apart, using 20 Hz stimulation. Followup visits will occur at 1, 4, and 12 weeks after both courses of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Are voluntary and competent to consent to treatment.
* Have met DSM-5 diagnostic criteria for borderline personality disorder, AND
* Have met DSM-5 diagnostic criteria of MDD single or recurrent, or Bipolar Disorder with a current Major Depressive Episode at the time of their consultation for rTMS.
* Are females between the ages of 18 and 65
* have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score of > 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF 1 or 2)
* have a score ≥18 on the HRSD-17 item
* able to adhere to the treatment schedule
* pass the TMS safety-screening questionnaire
* have normal thyroid functioning and no clinically significant abnormalities on CBC, on pre-study blood work.
* are already under the care of a psychiatrist who agrees to provide continuity of all non-rTMS aspects of care throughout the study.

Exclusion Criteria:

* Pregnancy
* A lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
* A MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, assessed by a study investigator to be primary and causing greater impairment than current MDDcurrent MDD or BPD
* Have received rTMS for any previous indication due to the potential compromise of subject blinding
* Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes.
* Have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth that cannot be safely removed
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
* Medication: currently (or in the last 4 weeks) taking more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy. Medication regimen should be stable for at least 4 weeks prior to first rTMS treatment.
* Alcohol or substance use: severe substance use disorder (based on DSM-5 diagnostic criteria) assessed by the study investigator to be primary and causing greater impairment than MDD or BPD.
* Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
* Serious suicide attempt that necessitate medical intervention during the last 3 months.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
HRSD-17 change | baseline to first followup (1 week post treatment), 3 months post-treatment
  The change in the 17-item Hamilton Rating Scale for Depression from baseline to first followup (1 week post treatment) for period 1 and 2 of the treatment

SECONDARY OUTCOMES:
ZAN-BPD change | baseline to first followup (1 week post treatment), 3 months post-treatment
  The change in the Zanarini Rating Scale for Borderline Personality Disorder from baseline to first followup (1 week post treatment) for period 1 and 2 of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jonathan Downar, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided